CLINICAL TRIAL: NCT01880216
Title: A Multinational, Multicentre, Randomized, Open, Parallel Group Study on the Efficacy and Safety of Bemiparin Sodium (LMWH) Compared to Enoxaparin Sodium (LMWH) in the Treatment of Acute Deep Vein Thrombosis (DVT)
Brief Title: Efficacy of Bemiparin Versus Enoxaparin in the Treatment of DVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bemiparin
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; DVT; Treatment; Low molecular weight heparin; Bemiparin; Enoxaparin
MeSH Terms: conditions — Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight; enoxaparin sodium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin sodium (Active Comparator): subcutaneous for 7±2 days and starting on Day 2 additionally the oral anticoagulant warfarin
  Interventions: Drug: Enoxaparin sodium
- Bemiprin sodium (Experimental): Bemiparin sodium (LMWH) s.c. for 7±2 days and starting on Day 2 additionally the oral anticoagulant warfarin
  Interventions: Drug: Bemiparin sodium

INTERVENTIONS:
Drug: Bemiparin sodium — subcutaneous application daily for 7±2 days
  Other Names: LMWH; CAS 874-98-4
  Arms: Bemiprin sodium
Drug: Enoxaparin sodium — subcutaneous for 7±2 days
  Other Names: LMWH; CAS 73334-07-3
  Arms: Enoxaparin sodium

SUMMARY:
Deep-vein thrombosis (DVT) is a common but under-diagnosed medical condition that occurs when a thrombus forms in one of the large veins, usually in the lower limbs, leading to either partial or complete blocked circulation. The condition may progress to severe health complications, such as pulmonary embolism (PE), if not diagnosed and treated in a timely and effective manner.

The goal of the therapy for lower-extremity DVT is to prevent the extension of thrombus and pulmonary embolism in the short term and to prevent recurrent events in the long-term. Although anticoagulant therapy decreases the risk of recurrent thrombosis, the treatment also increases the risk for major hemorrhage.

This trial aims to optimize the current medical knowledge on the effectiveness and safety of two low molecular weight heparins, bemiparin and enoxaparin in the treatment of deep vein thrombosis.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the therapeutic non-inferiority of bemiparin sodium (LMWH) versus enoxaparin sodium (LMWH) during a 7±2 days treatment period and a follow up of 11 weeks observation period.

Primary endpoint:

The percentage of patients with an improvement in thrombotic burden at Visit 3 (Day 83) defined as a ≥4-point reduction in thrombus score (or at least halving the thrombus score, when the total score is ≤ 6), without confirmed symptomatic extension of recurrence of DVT, confirmed symptomatic PE, or VTE-related death at Visit 3 (Day 83 / Month 3), as measured by complete compression ultrasound (cCUS) by Duplex sonography according to a standardized protocol.

Secondary endpoint:

The secondary efficacy endpoints are defined as the:

• Incidence of symptomatic venous thromboembolic events (VTE) at Visit 3 (Day 83:

* Recurrent DVT
* Pulmonary embolism

Incusion criteria:

Patients with acute deep-vein thrombosis of the leg (DVT) with symptoms of less than 14 days, confirmed by complete compression ultrasound (cCUS) within 48 hours prior study start.

Patients who have given their signed declaration of consent and data protection declaration Males and females aged 18 years

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute deep-vein thrombosis of the leg (DVT) with symptoms of less than 14 days confirmed by complete compression ultrasound (cCUS) within 48 h prior study starting .
2. Males and females aged ≥18 years
3. Patients who have given their written informed consent.

Exclusion Criteria:

Specific

1. History and presence of familial bleeding diathesis, presence of active bleeding contraindicating anticoagulant therapy, as well as presence of clinically relevant coagulation - and clotting factor disorder,and thrombocytopenia
2. Patients having undergone thrombectomy, having had insertion of a caval filter or who were treated with a fibrinolytic agent to treat the current episode of DVT
3. Treatment with heparin (fractionated or unfractionated), fondaparinux or vitamin K antagonist or warfarin for treatment of DVT for more than 48 h prior to enrolment
4. Long-term treatment with vitamin K antagonists, i.e. for atrial fibrillation, myocardial infarction or cardiomyopathy
5. Isolated distal calf vein thrombosis
6. Isolated superficial vein thrombosis
7. Any other symptomatic venous thromboembolism beside of DVT
8. Known hypersensitivity to heparin (including other pig-derived substances), to the study medications and heparin-derivatives including other LMWHs, warfarin and/or to the active ingredient or any excipient of the study medications
9. Concurrent treatment with platelet function inhibitors (such as acetylsalicylic acid, ticlopidine, clopidogrel, NSAID), fibrinolytic agents and other anticoagulant agents, Glycoprotein IIb/IIIa receptor- antagonists, nitro-glycerine iv, systemic glucocorticoids, penicillin in high doses, dextran, ascorbic acid, digitalis, tetracycline, medical products that could increase the potassium plasma level
10. History of documented or suspected heparin-induced thrombocytopenia (HIT I and II) or platelet count less than 100,000 platelets per mm3
11. Ischaemic stroke one month prior to enrolment
12. History of or active intracranial disorder (cerebral vascular aneurysm, arterio-venous malformation or cerebral neoplasm), history of haemorrhagic stroke or other intracranial bleeding 6 months prior to enrolment, active haemorrhage or increased risk of bleeding due to impaired haemostatics or organ lesion (e.g. peptic ulcer, hepatic failure, haemorrhagic stroke, macroscopic visible urogenital bleeding, cerebral vascular aneurysm or cerebral neoplasm) 1 month prior to enrolment.
13. Uncontrolled arterial hypertension: systolic blood pressure > 200 mmHg and diastolic blood pressure > 105 mmHg.
14. Severe impairment of pancreas function, history of gastro-duodenal ulcer disease, nephrolithiasis and/or ureterolithiasis, choroid and retinal vascular disease, suspected vascular retinopathy, vitreous haemorrhage or other intraocular bleedings, or any organic lesion with an increased risk of bleeding.
15. Significant liver disease (e.g. acute hepatitis, chronic active hepatitis, hepatic cirrhosis, hepatic encephalopathy) or liver enzymes (ALT and/or AST) > 5x ULN.

and others

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with an improvement in thrombotic burden at Visit 3 | 83±7 days

SECONDARY OUTCOMES:
Incidence of symptomatic venous thromboembolic events (VTE) | 83±7 days

OTHER OUTCOMES:
Treatment emergent adverse events (TEAEs) | 83±7 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Th Kaltwasser, Dr., Study Chair — Berlin-Chemie AG
Locations (25):
- Georgia (5):
  - Unimed Ajara LLC, Batumi
  - Angiology and Vascular Surgery Academic Clinic, Tbilisi
  - Bokhua Clinic of Angiology and Heart Diseases, Tbilisi
  - G. Chapidze Emergency Cardiology Centre, Tbilisi
  - Aversi Clinic, Tbilisi
- Russia (20):
  - Regional State Budget Institution of Healthcare "Regional Clinical Hospital", Barnaul
  - Federal State Budgetary Institution "Scientific Center of Reconstructive and Restorative Surgery" under Siberian Branch of the Russian Academy of Medical Sciences on the clinical base of State Institution of Healthcare, Irkutsk Regional Clinical Hospital, Irkutsk
  - State Healthcare Institution "Republican Clinical hospital of the ministry of Health of Republic Tatarstan, Kazan'
  - State Budget Public Health Institution of Moscow "City Clinical Hospital # 1 n.a. N.I. Pirogov", Moscow
  - Federal Government Healthcare Institution "Hospital of the Russian Federation Internal Affairs Ministry in Moscow", Moscow
  - Federally Funded State Institution "Institute of Surgery n.a. A.V. Vishnevskiy of the Ministry of Healthcare of Russian Federation", Moscow
  - State-Financed Healthcare Institution of the Novosibirsk Region "City Clinical Hospital # 2", Novosibirsk
  - State Budgetary Institution of the Omsk Region "Regional Clinical Hospital", Omsk
  - State Independent Healthcare Institution of the Perm kray "City Clinical Hospital # 4", Perm
  - State Budget Institution of Hifger Professional Education "Rostov State Medical University" of the Ministry of the Russian Federation, Rostov-on-Don
  - State Budgetary Institution of the Ryazan Region "Regional Clinical Cardiologic Dispensary", Ryazan
  - State Budget Institution "St.Petersburg Janelidze Research Institute of Emergency Medicine", Saint Petersburg
  - St. Petersburg State Public Health Institution "City Multi-field Hospital #2", Saint Petersburg
  - Nongovernmental Public Health Institution " Road Clinical Hospital" of Russian Railways, Saint Petersburg
  - State Educational Institution of Additional Professional Education "St.Petersburg Medical Academy of Postgraduate Education of Federal Agency for Health Care and Social Development", Chair of cardiovascular surgery, Saint Petersburg
  - St. Petersburg State Public Health Institution "City Hospital #26", Saint Petersburg
  - Federal State Budgetary Institution "Russian Center of Emergency and Radiation Medicine n.a. A.M. Nikiforov" of the Ministry of Russian Federation for Civil Defence, Emergencies and Elimination of Consequences of Natural Disasters, Saint Petersburg
  - State budgetary institution of higher professional education "Samara State Medical University", Samara
  - State Budget Public Health Institution of Yaroslavl region "Clinical hospital #10", Municipal Clinical Public Health Institution " Medical Unit of Novo-Yaroslavl Petroleum Refinery", Yaroslavl
  - State Budget Public Health Institution of Yaroslavl Region "Regional Clinical Hospital", Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suchkov IA, Martinez-Gonzalez J, Schellong SM, Garbade T, Falciani M; Bemiparin DVT Study Group. Comparison of Once-Daily Bemiparin with Twice-Daily Enoxaparin for Acute Deep Vein Thrombosis: A Multicenter, Open-Label, Randomized Controlled Trial. Clin Drug Investig. 2018 Feb;38(2):181-189. doi: 10.1007/s40261-017-0600-6. PMID 29214507